CLINICAL TRIAL: NCT05299320
Title: Covid 19 and Postural Sway: A Comprasion of SARS-CoV-2 and Healthy Sedentary Women
Brief Title: Postural Control in Covid-19
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Hikmet Kocaman, Head of study Dr. Hikmet Kocaman, Karamanoğlu Mehmetbey University
Other Study IDs: 12-2022/15
Record Dates: First submitted 2022-03-25; First posted 2022-03-29 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Performance
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Post-Covid: Being between the ages of 18-30, - Being a volunteer - Having had Covid-19 in the last 3 month Exclusion Criteria - Presence of neurologic and oncologic disease - Presence of orthopedic surgery - Presence of active Covid-19 disease - Any cardiopulmonary disease
  Interventions: Diagnostic Test: Neuromuscular fatigue and postural sway evaluation
- Healthy Person: Being between the ages of 18-30, Being a volunteer, not having Covid-19 before
  Interventions: Diagnostic Test: Neuromuscular fatigue and postural sway evaluation

INTERVENTIONS:
Diagnostic Test: Neuromuscular fatigue and postural sway evaluation — Neuromuscular fatigue will be established by using the Excalibur Sport Ergometer device and the Wingate Anaerobic Strength Test. Postural sway will be evaluated with Cyst Force Plate Balance device. This device is a precision device that provides objective measurable data.
  Other Names: Postural sway; Postural sway evaluation

SUMMARY:
This study was planned to investigate how much the anaerobic performance of individuals who experienced fatigue with Want (Wingate) affected their postural sway parameters.

DETAILED DESCRIPTION:
The postural sway parameters of the individuals will be evaluated using the "Kistler Force Plate" and the anaerobic values will be evaluated using the Wingate Anaerobic Strength Test and the "Excalibur Sport Ergometer" device. The data obtained will be compared with the data of patients with and without Covid-19 disease using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30, - Being a volunteer - Having had Covid 19 in the last 3 month

Exclusion Criteria:

* Presence of neurologic and oncologic disease - Presence of orthopedic surgery - Presence of active Covid 19 disease - Any cardiopulmonary disease

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with covid-19 and Have not had covid 19 before
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Postural Sway | 3 months
  Postural sway will be evaluated with Cyst Force Plate Balance device. This device is a precision device that provides objectively measurable data. Thanks to its movable platform, it can measure in all directions. Participants will be asked to stand on the platform assessing their body oscillations. They will be asked to look at a still picture on the wall with their arms at the iliac and eyes directly opposite them. Individuals will be asked to keep their designated positions for 30 seconds. At the end of the specified period, the data obtained from the device will be saved. Before and after the neuromuscular fatigue test postural sway will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Gökşen, PhD, Study Chair — Tarsus Universty
Locations (2):
- Turkey (Türkiye) (2):
  - Karamanoglu Mehmetbey University, Karaman
  - Karamanoğlu Mehmetbey University, Karaman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530